CLINICAL TRIAL: NCT06454305
Title: Comparative Effects of Active Cycle of Breathing Technique and Blow Bottle Technique to Prevent Post-operative Pulmonary Complications in Patients With Abdominal Surgeries Under General Anesthesia
Brief Title: Effects of ACBT and Blow Bottle Technique in Patients With Abdominal Surgeries Under General Anesthesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0380
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Abdominal Surgery
Keywords: Abdominal Surgeries; Active cycle of breathing Technique; Blow Bottle Technique; Pulmonary Complications,

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active cycle of breathing technique (Experimental): Breathing control, thoracic expansion and forced expiratory training are the three components of ACBT. The purpose of the thoracic expansion phase is to facilitate the release of secretions, enhance ventilation, and supply the necessary volume for forced expiratory breathing
  Interventions: Other: Active cycle of breathing technique
- Blow Bottle Technique (Active Comparator): 1-liter plastic bottle was filled with water to a height of 10 centimeters for this intervention. The water in the bottle was filled using a 30-cm-long tube that was placed 8 cm down. The participants were instructed to sit on a bed with comfortable position, Hold the bottle with one hand and the tube with the other Blowing Technique, Put the tube in mouth by holding lips firmly,Breathing in through nose and out through mouth,Blowing enough water is bubbled,Short Breaks for 2 to 3 mints, When mucus rises up get out of by cough and huff
  Interventions: Other: Blow Bottle Technique

INTERVENTIONS:
Other: Active cycle of breathing technique — Breathing control, thoracic expansion and forced expiratory training are the three components of ACBT. The purpose of the thoracic expansion phase is to facilitate the release of secretions, enhance ventilation, and supply the necessary volume for forced expiratory breathing. Secretions are moved into the central airways during the forceful expiratory exercise that follows The three stages of ACBT
  Arms: Active cycle of breathing technique
Other: Blow Bottle Technique — A 1-liter plastic bottle was filled with water to a height of 10 centimeters for this intervention. The water in the bottle was filled using a 30-cm-long tube that was placed 8 cm down. The participants were instructed to sit on a bed with comfortable position, Hold the bottle with one hand and the tube with the other Blowing Technique, Put the tube in mouth by holding lips firmly, Breath in through nose and out through mouth, Blowing enough water is bubbled, Short Breaks for 2 to 3 mints, When mucus rises up get out of it by coughing or huffing
  Arms: Blow Bottle Technique

SUMMARY:
A postoperative pulmonary complication (PPC) is the most common serious complication after Abdominal surgery under GA which lead to longer hospital stays and have deleterious outcomes on lung volumes, mucociliary clearance, accumulation of mucus, saliva and cough reflex. Chest physiotherapy for airway clearance which includes postural drainage, chest percussion, vibrations, Along with these, breathing exercises such ACBT and Blow bottle technique are recommended to clear secretion which aid in enhancing pulmonary function by effectively mobilizing and eliminating excess bronchial secretions.

This study of randomized clinical trial will check the comparative effect of ACBT and Blow Bottle Technique in patients with abdominal surgeries under GA by taking a sample of 44 patients through non probability convenience sampling technique. Subject of both gender will be included between the age of 30 to 50 years who will undergoes with elective abdominal surgeries under GA (Cholecystectomy, Hysterectomy ,Appendectomy, Hemorrhoidectomy) and Laparoscopic /open. Elective surgeries under spinal anesthesia, emergency surgeries, cardiothoracic surgeries and hemodynamically unstable subjects will be excluded. 22 subjects will receive ACBT and other 22 subjects will receive Blow bottle technique for 20 minutes duration per session, two sessions per day for a period of 5 days. The status of airway clearance, oxygen saturation and lungs volumes will be measured pre and post intervention on day 1 and at the end of 5th day by using BCSS, Pulse oximeter and Spirometer.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 to 50 Gender: male/Female Both Elective surgeries Under General Anesthesia (Cholecystectomy, Hysterectomy ,Appendectomy, Hemorrhoidectomy) Laparoscopic /open both POCs: Sputum retention, hypoxemia, impair pulmonary function From the day 0 or immediate after surgery

Exclusion Criteria:

* Elective surgeries under spinal anesthesia Emergency surgeries Cardiothoracic surgeries Neurological impairment, prolong surgeries Psychological impairment Head and neck surgeries and vascular surgeries Hemodynamically unstable

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Pulse Oximeter | baseline and fourth week
  An invasive technique for keeping an eye on someone's blood oxygen saturation is pulse oximetry. The accuracy of peripheral oxygen saturation measurements is usually 2% of the arterial oxygen saturation level obtained from arterial blood gas analysis, which is a more precise measurement. It may decrease and remain low owing to specific cardiovascular problems, or it may peak and climb after a run or other physical activity. Nonetheless, conventional research indicates that the usual range for pulse rate on an oximeter in healthy persons is between 60 and 100 beats per minute
Spirometer | baseline and fourth week
  The most used pulmonary function test is spirometry. It assesses the capacity of the lungs to breathe in and out, especially the volume and/or velocity of air that can be expelled. When evaluating breathing patterns to detect diseases including asthma, pulmonary fibrosis, cystic fibrosis, and COPD, spirometry is useful. An FEV1/FVC ratio larger than 0.70 with both FEV1 and FVC over 80% of the expected value are considered normal spirometry data. TLC exceeding 80% of the predicted value is typical in the event that lung volumes are measured. Diffusion capacity that is more than 75% of the expected value is likewise regarded as typical
Breathlessness, Cough and Sputum Scale (BCSS) | baseline and fourth week
  A three-item questionnaire used to evaluate the patient's cough, sputum, and dyspnea forms the basis of the BCSS. Using a Likert scale, with 0 denoting improved symptoms and a 4 denoting deteriorating symptoms, individuals can register their symptoms on the BCSS. Patients are asked to assess the severity of each of the three symptoms on a 5-point scale as part of the BCSS, a patient-reported outcome measure. Higher scores denote more severe symptoms. A total score is obtained by adding the item scores

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Afzal, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Cairns Railway Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cui Y, Cao R, Li G, Gong T, Ou Y, Huang J. The effect of lung recruitment maneuvers on post-operative pulmonary complications for patients undergoing general anesthesia: A meta-analysis. PLoS One. 2019 May 29;14(5):e0217405. doi: 10.1371/journal.pone.0217405. eCollection 2019. PMID 31141541
- [Background] Kokotovic D, Berkfors A, Gogenur I, Ekeloef S, Burcharth J. The effect of postoperative respiratory and mobilization interventions on postoperative complications following abdominal surgery: a systematic review and meta-analysis. Eur J Trauma Emerg Surg. 2021 Aug;47(4):975-990. doi: 10.1007/s00068-020-01522-x. Epub 2020 Oct 7. PMID 33026459
- [Background] Boden I, Robertson IK, Neil A, Reeve J, Palmer AJ, Skinner EH, Browning L, Anderson L, Hill C, Story D, Denehy L. Preoperative physiotherapy is cost-effective for preventing pulmonary complications after major abdominal surgery: a health economic analysis of a multicentre randomised trial. J Physiother. 2020 Jul;66(3):180-187. doi: 10.1016/j.jphys.2020.06.005. Epub 2020 Jul 14. PMID 32680742